CLINICAL TRIAL: NCT04496141
Title: Evaluation of Commercial SARS-CoV-2 Antibody Immunoassays for COVID-19
Status: Completed | Type: Observational
Sponsor: Hong Kong Sanatorium & Hospital (Industry)
Responsible Party: Principal Investigator, Dr. Jonpaul ST Zee, Specialist in Infectious Disease, Hong Kong Sanatorium & Hospital
Other Study IDs: RC-2020-12
Record Dates: First submitted 2020-07-30; First posted 2020-08-03 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- With COVID-19 infection: Subjects with a positive SARS-CoV-2 PCR
  Interventions: Diagnostic Test: SARS-CoV-2 antibody immunoassays
- Without COVID-19 infection: Subjects with COVID-19 negative serum
  Interventions: Diagnostic Test: SARS-CoV-2 antibody immunoassays

INTERVENTIONS:
Diagnostic Test: SARS-CoV-2 antibody immunoassays — Different commercial SARS-CoV-2 antibody immunoassays

SUMMARY:
Achieved serum samples of persons with or without evidence of COVID-19 infection are tested using the different commercial SARS-CoV-2 antibody immunoassays. The performance of the immunoassays is then assessed by comparing the 2 groups of samples.

DETAILED DESCRIPTION:
Achieved serum samples of the different testing groups are retrieved and tested with the immunoassays according to manufacturer's instruction.

The test results are then compared and analyzed with statistical tests to assess the immunoassays'performance

ELIGIBILITY:
Inclusion criteria for COVID-19 infected sera: any patient with PCR confirmed COVID-19 infection

Inclusion criteria for COVID-19 negative sera: sera collected after a negative SARS-CoV-2 PCR

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who attended clinic and had a positive SARS-CoV-2 PCR and subjects who had COVID-19 negative serum during the epidemic in Hong Kong.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
The accuracy of the different commercial SARS-CoV-2 antibody immunoassays | 1 month
  To investigate the accuracy (including sensitivity, specificity, positive and negative predictive value) of the commercial SARS-CoV-2 antibody immunoassays

CONTACTS AND LOCATIONS:
Overall Officials: Jonpaul Sze Tsing Zee, MBChB, Principal Investigator — Hong Kong Sanatorium & Hospital
Locations (1):
- Hong Kong Sanatorium & Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No